CLINICAL TRIAL: NCT07144098
Title: Study of Pharmacokinetics and Safety of GZR18 Injection in Subjects With Liver Insufficiency and Normal Liver Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GZR18-BWM-107
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Obesity/Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GZR18 injection (Experimental)
  Interventions: Drug: GZR18 injection

INTERVENTIONS:
Drug: GZR18 injection — 3 mg-Control group
Drug: GZR18 injection — 3 mg-mild liver insufficiency
Drug: GZR18 injection — 3 mg-moderate liver insufficiency
Drug: GZR18 injection — 3 mg-severe liver insufficiency

SUMMARY:
This study adopts a multicenter, single-dose, open-label, and parallel design, which is aimed at assessing the PK and safety profiles of GZR18 Injection in subjects with normal liver function and those with mild, moderate or severe liver insufficiency.

The study duration for each subject in this study is up to 50 days, including a screening period of up to 14 days (Day-14 to Day-1), an 8-day dosing/observation period (Day 1 to Day 8), and a 28-day follow-up period (Day 9 to Day 36).

ELIGIBILITY:
Inclusion Criteria:

* All Subjects:

  1. Subjects who fully understand the study contents, study procedures and possible risks, can follow the contraindications and restrictions specified in this protocol, and voluntarily sign the informed consent form.
  2. Subjects (male or female) age ≥ 18 and ≤ 75 years at the time of signing the ICF.
  3. Weight ≥ 50 kg for males and ≥ 45 kg for females, with a body mass index (BMI) of 19.0-32.0 kg/m2 (both inclusive).
  4. Subjects with childbearing potential from signing the ICF to 8 weeks after the last dose have no family planning, are willing to adopt effective contraceptive measures and have no plans for sperm donation or egg donation; women of childbearing potential are not pregnant or lactating: they must have a negative pregnancy test at screening and have no unprotected sexual intercourse within 2 weeks before screening.

     Only for Subjects with Liver Dysfunction:
  5. Chronic liver insufficiency caused by viral hepatitis, alcoholic liver disease, autoimmune hepatitis or other reasons, and after comprehensive assessment by researchers, the disease is not in the rapid progression stage.
  6. Determined as grade A, B or C according to the Child-Pugh score, and no albumin was used within 21 days before screening.
  7. Researchers determine the physical condition of those who are eligible for this test based on medical history inquiry, physical examination, vital signs, clinical laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine, etc.), 12-lead electrocardiogram, chest X-ray, B-ultrasound, etc.

Only for Subjects with Normal Liver Function:

1. Matched with the subjects in the liver insufficiency group in terms of mean age (±10 years), sex ±1, mean weight (±10 kg), and mean BMI (±20%).
2. Those whose clinical laboratory tests, vital signs, physical examinations, electrocardiograms, chest X-rays, B-ultrasound and other tests are normal, or who are evaluated as abnormal by the researcher but have no clinical significance.

Exclusion Criteria:

* 1. Subjects with an allergic constitution, including those with a history of severe drug hypersensitivity or allergy, and known to be allergic to the investigational drug or GLP-1 drugs or any component in the investigational drug (citrate, sodium chloride, disodium hydrogen phosphate, hydrochloric acid and sodium hydroxide).

  2. History of acute or chronic pancreatitis and pancreatic injury before screening. Subjects with symptomatic gallbladder disorders at screening.

  3. History or relevant family history of medullary thyroid carcinoma, multiple endocrine neoplasia (MEN) 2A or 2B before screening.

  4. Have the following cardiovascular and cerebrovascular diseases within 6 months before screening: Decompensated cardiac insufficiency (New York Heart Association NYHA Class III or IV), angina unstable or myocardial infarction, history of heart valve replacement surgery, coronary artery bypass grafting or other invasive cardiovascular surgery including percutaneous coronary intervention, ischemic or hemorrhagic stroke (excluding lacunar infarction), or transient ischemic attack.

  5. During screening, 12-lead electrocardiogram: QTcF > 470 msec (for males) or > 480 msec (for females).

  6. Those with a history of severe active infection within one month prior to screening.

  7. Subjects with a history of malignant tumors within the past 5 years (except for basal cell carcinoma of ski, squamous cell carcinoma of skin or in situ cancer of cervix).

  8. Subjects with severe trauma, gastrointestinal surgery, or other major surgical operations within 4 weeks before screening.

  9. Subjects who are unwilling or unable to comply with the study procedures specified in the protocol, or who are deemed unsuitable for participating in this clinical study by any investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-07-12 (Estimated); Study Completion 2027-01-26 (Estimated)

PRIMARY OUTCOMES:
Cmax:Maximum plasma concentration. | through study completion, an average of 36 days
AUC0-last:Area under the plasma concentration-time curve at 0 h to last observation time-point after a single dose. | through study completion, an average of 36 days
AUC0-inf:Area under the plasma concentration-time curve at 0 h to infinity after a single dose. | through study completion, an average of 36 days

SECONDARY OUTCOMES:
AUC0-336 h：Area under the plasma concentration-time curve from time zero to 336 hours | through study completion, an average of 36 days
Tmax:Time of Maximum Drug ConcentrationTime to Maximum aentration | through study completion, an average of 36 days
TEAE：Treatment Emergent Adverse Event | through study completion, an average of 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Liyuan Zhao Ph.D, Study Director — Gan & Lee Pharmaceuticals.
Locations (1):
- Gan & Lee Pharmaceuticals, Beijing, China